CLINICAL TRIAL: NCT03548324
Title: Enteral Nutrition Tolerance and Non-invasive Respiratory Support in Preterm Infants
Brief Title: Enteral Nutrition Tolerance And REspiratory Support (ENTARES)
Acronym: ENTARES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Cresi, MD, PhD, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENTARES
Record Dates: First submitted 2018-04-28; First posted 2018-06-07 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Very Low Birth Weight Infant; Respiratory Distress Syndrome in Premature Infant; Enteral Feeding Intolerance
Keywords: Feeding Tolerance; RDS; HFNC; NCPAP; Preterm; NEC; Enteral Nutrition; Non Invasive Respiratory Support; Very Low Birth Weight Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Two arms multicenter randomized controlled trial designed according to the intention-to-treat model. The assignement to one of the two arms (NCPAP or HHHFNC) is by block randomization. The randomization program is designed to obtain, in each research unit, a balance between the two arms according to gestation age (GA <28 weeks and GA ≥ 28 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHHFNC (Active Comparator): Heated Humidified High Flow Nasal Cannulae
  Interventions: Device: HHHFNC
- NCPAP (Active Comparator): Nasal Continuous Positive Air Pressure
  Interventions: Device: NCPAP

INTERVENTIONS:
Device: HHHFNC — Application to HHHFNC to treat respiratory distress syndrome in preterm infants previously demonstrated to be stable on a non-invasive respiratory support (HHHFNC or NCPAP).
  Arms: HHHFNC
Device: NCPAP — Application to NCPAP to treat respiratory distress syndrome in preterm infants previously demonstrated to be stable on a non-invasive respiratory support (HHHFNC or NCPAP).
  Arms: NCPAP

SUMMARY:
This research study aims to evaluate the relation between non-invasive ventilation and feeding tolerance in preterms with respiratory distress syndrome (RDS).

To this purpose a multicenter randomized controlled trial was designed. It will involve 13 neonatal intensive care units (NICUs) in Italy and will be coordinated by the NICU of the University of Turin.

The study focuses on the impact of two non-invasive respiratory support techniques (NCPAP and HHHFNC) on feeding intolerance and gastrointestinal complications to identify which technique is the most effective and safe in preterms with RDS. Further aim is to identify which technique could be the most suitable for full enteral feeding achievement and acquisition of oral feeding. Improving enteral feeding tolerance and promoting oral feeding could improve clinical outcomes and reduce risks and costs of prolonged hospital stay.

Further aim is to evaluate the response to NCPAP and HHHFNC in the treatment of RDS, focusing on a population of extremely low preterms.

DETAILED DESCRIPTION:
BACKGROUND:

Respiratory distress syndrome (RDS) is a common condition in premature infants and one of the major cause of neonatal mortality. For many years, preterm infants with RDS have been treated with mechanical ventilation increasing risks of acute lung injury and long-term morbidity, as bronchopulmonary dysplasia (BPD). Early nasal continuous positive airway pressure (NCPAP) treatment combined with surfactant replacement therapy decreases the need for mechanical ventilation and has been recommended as first line treatment for RDS. However, NCPAP has significant limitations, mainly related to the type of interface needed. Excessive leak around the prongs or mask and through the mouth can lead to inadequate support, whereas excessive pressure may result in pneumothorax and damage of the nose and face. Moreover, the bulky fixation devices obscure the infant's face both interfering with feeding and positioning. In recent years, heated humidified high-flow nasal cannula (HHHFNC) has been studied as an alternative non-invasive respiratory supports (NIReS). HHHFNC became popular partially thanks to some perceived advantages related to the type of interface used. Cannulae are easier to apply than NCPAP prongs or mask, may be more comfortable for infants, and may enable easier access to babies' faces, thus facilitating feeding and parental bonding. Whereas practical advantages seem to be established there is controversy about HHHFNC efficacy as respiratory support. Recent studies support that HHHFNC is as effective as NCPAP for the primary treatment of RDS, but evidences are still insufficient and data are still lacking, especially for the extremely preterm population (<28 weeks of gestation). A recent Cochrane comparing HHHFNC with other NIReS showed equivalent rates of treatment failure and similar rates of BPD when used as a post-extubation support in preterm infants. With equivalent effectiveness, the choice of the most adequate NIReS should consider the impact on the health status of the premature evaluating, above all, the effect on nutrition and growth. Along with RDS, feeding intolerance (FI) represents a relevant issue in preterm infants and the coexistence of the two represents a great challenge for the neonatologist. Because of gastrointestinal immaturity, almost 1:3 preterm infants develops clinical symptoms of FI causing interruptions of feeding which delays the establishment of adequate enteral nutrition and prolongs the need for parental nutrition thus increasing the risk of infections and prolonging hospital stay. Avoiding FI and its complication, as necrotizing enterocolitis (NEC), is a priority for the neonatologist, who often faces the challenge of interpreting the clinical and prognostic significance of common and aspecific signs of FI. Clear identification of the parameters that should be evaluated to identify FI is still lacking in literature, although, among controversy, the presence of gastric residuals, vomits and/or regurgitations, abdominal distension and the onset of crises of apnea/bradycardia are considered the most frequent signs. Literature and clinical practise suggest that a correlation between non-invasive ventilation and the occurrence of FI and NEC exists even if the mechanisms through which ventilation may induce FI and its incidence in ventilated infants are still unclear. Considering NIReS, the most common hypothesis is that pressurized gasses, that are not completely conveyed to the airways, could cause bowel distension. Bowel distension in infants on CPAP was described by Jaile et al. as CPAP belly syndrome but no inferences about feeding tolerance and risk of NEC was drawn. More recent studies evaluated the effect of CPAP on mesenteric flow and gastric emptying suggesting a role of CPAP as a risk factor for FI. No specific studies have been designed to evaluate the impact of different NIReS on FI and the occurrence of NEC, which are generally evaluated as secondary outcomes, susceptible to data analysis and patient selection biases. Our hypothesis is that different techniques of NIReS may have different impact on feeding issues in preterm infants. Therefore, our study will focus on the impact that the two most common NIReS (NCPAP and HHHFNC) have on feeding.

PROJECT AIMS AND DESIGN:

Aim of the study is to evaluate the effects on feeding tolerance of different NIReS techniques (NCPAP vs HHHFNC) in preterm infants with RDS and to evaluate their impact on full enteral feeding achievement and acquisition of oral feeding. Further aim is to evaluate the response to NCPAP and HHHFNC as treatment for RDS in extremely preterm infants. To these purposes a multicenter randomized controlled trial was designed. The research project will involve 13 neonatal intensive care units (NICU) in Italy and will be coordinated by the NICU of the University of Turin.

PATIENTS:

Basing on a population of infants with a gestational age <30 weeks and consecutively admitted to the NICUs of each research unit from January to June 2017 (mean time of FEF: 19.6 days, delta: 5.7) and considering a ratio between the subjects of the two arms of 1:1, the sample size to observe a difference of 30% between the 2 arms has been set at 141 patients per arm.

PROTOCOL:

After randomization each infant will be subsequently enrolled into the study and treated with NCPAP or HHHFNC as per randomization. Each research unit will refer to its own protocols for ventilation and nutrition, although respecting some minimal standard criteria and indications, common and approved by all research units. Common criteria for ventilation regard the suggested initial setup of NCPAP and HHHFNC and the indications suggested to try weaning and define failure and are listed below:

Suggested initial setup:

CPAP between 5 and 7 cmH2O if on NCPAP and flow between 4 and 7 L/min if on HHHFNC; FiO2 is set as to reach pO2 = 50 - 60 mmHg and SatO2 TC = 90 - 95%.

Criteria to try weaning:

CPAP < 4 cmH2O if on NCPAP and flow < 2 if on HHHFNC with FiO2 < 25% to maintain pO2 = 50 - 60 mmHg and SatO2 TC = 90 - 95%.

Failure criteria:

* FiO2 > 40%
* pH < 7.2
* pCO2 > 65 mmHg
* ≥ 3 episodes of desaturations (SatO2 TC ≤ 80%) per hour
* ≥ 3 episodes of apnea (> 20 sec) and/or bradycardia (FC ≤ 80 bpm) per hour
* Silverman score > 6

The indications for the interruption of feeding are based on abdominal examination, on the occurrence of vomits/regurgitations and crises of apnea/bradycardia and on the evaluation of alvus and gastric residual volumes, if required by the protocol of the unit. The maximum cut-off for feeding progression is set at 30 mL/Kg/day. Data on ventilation, nutrition, growth and clinical events will be collected from enrollment to discharge.

DATA ANALYSIS:

Data will be analysed according to an intention-to-treat model. Therefore, data from all infants enrolled into the study will be considered for the analysis. Death and transfer to another hospital, before reaching full enteral feeding, are the only two reasons for exclusion. The primary outcome will be evaluated by a survival analysis with non-parametric distribution. Secondary outcomes will be evaluated by Fisher's exact test or appropriate generalized linear models.

EXPECTED RESULTS AND IMPACT ON CLINICAL PRACTICE:

The identification of the most suitable NIReS for preterm infants with RDS and FI could reduce gastrointestinal complications, improve growth and reduce hospital stay, thus improving quality of life of infants and their family and reducing health costs. The evaluation of the timing of oral feeding could be useful to understand the influence that NIReS techniques have on the development of sucking-swallowing coordination. The evaluation of the response to NCPAP and HHHFNC could clarify their efficacy as treatment for RDS in extremely preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RDS
* stability on HHHFNC or NCPAP since at least 48 hours (SatO2 TC 90-95%, pCO2 ≤ 60 mmHg, FiO2 < 40%, Silverman score ≤ 6, ≤ 2 apnea episodes/hour with CPAP ≤ 7 cmH2O if on NCPAP and flow ≤ 6 L/min if on HHHFNC )
* ≤ 7 days of life
* suitability to start enteral feeding (if not already started)
* parental written consent

Exclusion Criteria:

* neurological or surgical diseases
* sepsis
* chromosomal abnormalities or major malformations

Ages: 25 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Full Enteral Feeding (FEF) time | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Time to reach Full Enteral Feeding, defined as an enteral intake of 150 mL/kg/die (n. of days)

SECONDARY OUTCOMES:
Half Enteral Feeding (HEF) time | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Time to reach Full Enteral Feeding/2, defined as an enteral intake of 75 mL/kg/die (n. of days)
Enteral feeding interruptions | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Median number of feeding interruptions per day
Not given feeds | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Median number of not given feeds per day
Pathologic gastric residuals | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Median number of pathologic gastric residuals per day
Vomits and/or regurgitations | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Median number of vomits and/or regurgitations per day
Abdominal distension | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Median abdominal distension score per day
Beginning of oral feeding | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Post-menstrual age when bottle- or breast-feeding is started
Full oral feeding time | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Post-menstrual age when full bottle- or breast-feeding is achieved
Weight growth | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Weight growth evaluated through Δ z-score analysis
Duration of respiratory support assigned at randomization | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Time during which the non-invasive respiratory support device assigned at randomization is maintained
Total duration of respiratory support need | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Time during which any kind of respiratory support is needed
Failure of the respiratory support assigned at randomization | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Failure of the respiratory support assigned and need for mechanical ventilation or different kind of respiratory support (n. of days)
Length of hospital stay | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Total duration of hospital stay (n. of days)
Complications | From date of randomization until the date of hospital discharge or date of death, whichever came first, assessed up to 6 months
  Occurrence of complications as NEC, bowel perforation, pneumothorax, BPD, retinopathy of the premature.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, MD, PhD, Study Director — Città della Salute e della Scienza, S.C. Neonatologia U., University of Turin
Locations (13):
- Italy (13):
  - AOUC Policlinico di Bari, Bari, Bari (BA)
  - ASL Ospedale Di Venere, Bari, Bari (BA)
  - Ospedale Sana Croce e Carle, Cuneo, CN
  - AOU Careggi, Florence, Firenze (FI)
  - ASST Grande Ospedale Metropolitano Niguarda, Milan, Milano (MI)
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico (Mangiagalli), Milan, Milano (MI)
  - Ospedale dei Bambini Vittore Buzzi, Milan, MI
  - AOU Federico II, Napoli, Napoli (NA)
  - Ospedale San Matteo, Pavia, PV
  - Fondazione Policlinico Universitario A. Gemelli, Roma, Roma (RM)
  - AOU Città della Salute e della Scienza di Torino - Ospedale S.Anna, Torino, Torino (TO)
  - AOU Città della Salute e della Scienza di Torino - Ospedale S.Anna, Torino, TO
  - ASST Sette Laghi Polo Universitario, Varese, Varese (VA)

REFERENCES:
- [Background] Davies PL, Maxwell NC, Kotecha S. The role of inflammation and infection in the development of chronic lung disease of prematurity. Adv Exp Med Biol. 2006;582:101-10. doi: 10.1007/0-387-33026-7_9. PMID 16802622
- [Background] Lista G, Maturana A, Moya FR. Achieving and maintaining lung volume in the preterm infant: from the first breath to the NICU. Eur J Pediatr. 2017 Oct;176(10):1287-1293. doi: 10.1007/s00431-017-2984-y. Epub 2017 Aug 10. PMID 28795220
- [Background] Aly H. Ventilation without tracheal intubation. Pediatrics. 2009 Aug;124(2):786-9. doi: 10.1542/peds.2009-0256. Epub 2009 Jul 27. No abstract available. PMID 19651592
- [Background] Ramanathan R, Sekar KC, Rasmussen M, Bhatia J, Soll RF. Nasal intermittent positive pressure ventilation after surfactant treatment for respiratory distress syndrome in preterm infants <30 weeks' gestation: a randomized, controlled trial. J Perinatol. 2012 May;32(5):336-43. doi: 10.1038/jp.2012.1. Epub 2012 Feb 2. PMID 22301528
- [Background] Fischer HS, Buhrer C. Avoiding endotracheal ventilation to prevent bronchopulmonary dysplasia: a meta-analysis. Pediatrics. 2013 Nov;132(5):e1351-60. doi: 10.1542/peds.2013-1880. Epub 2013 Oct 21. PMID 24144716
- [Background] Schmolzer GM, Kumar M, Pichler G, Aziz K, O'Reilly M, Cheung PY. Non-invasive versus invasive respiratory support in preterm infants at birth: systematic review and meta-analysis. BMJ. 2013 Oct 17;347:f5980. doi: 10.1136/bmj.f5980. PMID 24136633
- [Background] Wilkinson D, Andersen C, O'Donnell CP, De Paoli AG, Manley BJ. High flow nasal cannula for respiratory support in preterm infants. Cochrane Database Syst Rev. 2016 Feb 22;2(2):CD006405. doi: 10.1002/14651858.CD006405.pub3. PMID 26899543
- [Background] Kotecha SJ, Adappa R, Gupta N, Watkins WJ, Kotecha S, Chakraborty M. Safety and Efficacy of High-Flow Nasal Cannula Therapy in Preterm Infants: A Meta-analysis. Pediatrics. 2015 Sep;136(3):542-53. doi: 10.1542/peds.2015-0738. Epub 2015 Aug 17. PMID 26283781
- [Background] Yoder BA, Manley B, Collins C, Ives K, Kugelman A, Lavizzari A, McQueen M. Consensus approach to nasal high-flow therapy in neonates. J Perinatol. 2017 Jul;37(7):809-813. doi: 10.1038/jp.2017.24. Epub 2017 Mar 23. PMID 28333157
- [Background] Salvo V, Lista G, Lupo E, Ricotti A, Zimmermann LJI, Gavilanes AWD, Gitto E, Colivicchi M, Ferrau V, Gazzolo D. Comparison of three non-invasive ventilation strategies (NSIPPV/BiPAP/NCPAP) for RDS in VLBW infants. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2832-2838. doi: 10.1080/14767058.2017.1357693. Epub 2017 Aug 1. PMID 28718356
- [Background] Mihatsch WA, Pohlandt F, Franz AR, Flock F. Early feeding advancement in very low-birth-weight infants with intrauterine growth retardation and increased umbilical artery resistance. J Pediatr Gastroenterol Nutr. 2002 Aug;35(2):144-8. doi: 10.1097/00005176-200208000-00008. PMID 12187288
- [Background] Parker L, Torrazza RM, Li Y, Talaga E, Shuster J, Neu J. Aspiration and evaluation of gastric residuals in the neonatal intensive care unit: state of the science. J Perinat Neonatal Nurs. 2015 Jan-Mar;29(1):51-9; quiz E2. doi: 10.1097/JPN.0000000000000080. PMID 25633400
- [Background] Li YF, Lin HC, Torrazza RM, Parker L, Talaga E, Neu J. Gastric residual evaluation in preterm neonates: a useful monitoring technique or a hindrance? Pediatr Neonatol. 2014 Oct;55(5):335-40. doi: 10.1016/j.pedneo.2014.02.008. Epub 2014 Aug 14. PMID 25129325
- [Background] Gephart SM, Fleiner M, Kijewski A. The ConNECtion Between Abdominal Signs and Necrotizing Enterocolitis in Infants 501 to 1500 g. Adv Neonatal Care. 2017 Feb;17(1):53-64. doi: 10.1097/ANC.0000000000000345. PMID 27754992
- [Derived] Cresi F, Maggiora E, Lista G, Dani C, Borgione SM, Spada E, Ferroglio M, Bertino E, Coscia A; ENTARES Study Group. Effect of Nasal Continuous Positive Airway Pressure vs Heated Humidified High-Flow Nasal Cannula on Feeding Intolerance in Preterm Infants With Respiratory Distress Syndrome: The ENTARES Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2323052. doi: 10.1001/jamanetworkopen.2023.23052. PMID 37436750
- [Derived] Cresi F, Maggiora E, Borgione SM, Spada E, Coscia A, Bertino E, Meneghin F, Corvaglia LT, Ventura ML, Lista G; ENTARES Study Research Group. Enteral Nutrition Tolerance And REspiratory Support (ENTARES) Study in preterm infants: study protocol for a randomized controlled trial. Trials. 2019 Jan 18;20(1):67. doi: 10.1186/s13063-018-3119-0. PMID 30658676